CLINICAL TRIAL: NCT04415853
Title: Lerotinib Versus Investigator's Choice Single-agent Chemotherapy in Patients With Locally Advanced/Metastatic Esophageal Squamous Cell Carcinoma and EGFR Overexpression That Progressed After Second-line Therapy:Phase 3 Study
Brief Title: Study of Larotinib in Unresectable Advanced or Recurrent Esophageal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCD-DZ650-20-001
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Esophageal Cancer
Keywords: ESCC;; EGFR overexpression;; Phase 3
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Irinotecan; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lerotinib Arm (Experimental): 350 mg,qd, orally about half an hour after a meal, continuous administration, every 21 days for a treatment cycle.
  Interventions: Drug: Lerotinib
- Active Comparator Arm (Active Comparator): Irinotecan: Intravenously administered at a dose of 180 mg/m2 every 2 weeks until documented disease progression, discontinuation due to toxicity, withdrawal of consent or the study ends.
  Tegafur: 40-60mg po bid(d1-d14),every 21 days as a cycle, continuous drug administration from 1 to 14 days of each cycle, and then stopped 7 days.
  Interventions: Drug: Irinotecan/Tegafur

INTERVENTIONS:
Drug: Lerotinib — Specification: 50 mg/capsule and 150 mg/capsule
  Other Names: Z650
  Arms: Lerotinib Arm
Drug: Irinotecan/Tegafur — Irinotecan:Specification: 2mL: 40mg;5mL:0.1g Tegafur:20mg/capsule
  Other Names: Irinotecan Hydrochloride Injection/Tegafur Gimeracil Oteracil Potassium Capsule
  Arms: Active Comparator Arm

SUMMARY:
This is a randomized, controlled, multi-center, open trial, unresectable locally advanced or metastatic esophageal squamous cell carcinoma patients that failed at least second-line treatment and overexpressed EGFR were enrolled and randomly assigned to the experimental group and control group at a 1: 1 ratio.,who received Larotinib and the chemotherapy regimen chosen by the investigator (Irinotecan Hydrochloride Injection or Tegafur Gimeracil Oteracil Potassium Capsule),respecitively.

Subjects are administered until disease progression assessed by the RECIST V1.1 standard (unless the investigator evaluates that the subject continues to have clinical benefit from continuing treatment, the subject may be allowed to continue treatment), and begins to receive new anti-tumor treatment, unacceptable toxicity, withdrawal of informed consent, or other conditions that meet the criteria for terminating trial treatment / withdrawal from the trial.

The research phase of this study is divided into pre-screening period (~ D-28), screening period (D-28 ~ D-1), treatment period, treatment end visit (± 7 days after the last dose), safety follow-up ( Until 28 ± 7 days after the last dose) and survival follow-up.

DETAILED DESCRIPTION:
The experimental group and the control group were administered until the disease progression assessed by the RECIST V1.1 standard (unless The investigator evaluates that the subject continues to have clinical benefits, and the subject can be allowed to continue receiving treatment), start new anti-tumor therapy, unacceptable toxicity, withdraw informed consent, ect.

The research phase of this study is divided into screening period, treatment period, treatment end visit, safety follow-up and survival follow-up.

Subjects who have finished the screening examination and evaluation after the screening period enter the treatment period, and evaluate the efficacy. Subjects who have finished the treatment need to continue to undergo safety follow-up ; For subjects who have finished the trial treatment due to toxic reactions or other reasons, and have not observed the progression, they still need to carry out imaging evaluation according to the original frequency until the occurrence of tumor progression judged by RECIST V1.1 standard, start of new anti-tumor therapy, withdrawal of informed consent, loss of follow-up, death, or end of study, whichever occurs first; all subjects receive survival follow-up until death,lost of ,the follow-up or the study ended，whichever occurred first.

PK studies: Pharmacokinetic (PK) studies are conducted only in centers with appropriate conditions. Only some subjects in the experiemtal group are required to undergo a PK study. Participate in intensive PK blood collection (8-12 cases), and participate in sparse PK blood collection (150 cases). Subjects participating in intensive PK blood collection do not participate in sparse PK blood collection.

Biomarker research: Detect EGFR overexpression and amplification research on tumor tissue samples for all subjects and explore the relationship between its efficacy and changes in EGFR overexpression and amplification status before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-75 years, male or female.
2. Histologically or cytologically confirmed squamous cell carcinoma of the esophagus or advanced/metastatic disease.
3. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Life expectancy of greater than 3 months.
5. Documented objective radiographic or clinical disease progression on two previous lines of standard therapy.
6. Can provide archival tumor tissue sample for biomarker analysis (such as EGFR overexpression/expansion status), biopsies are required if tissue samples cannot be provided
7. Confirmed by the central laboratory as EGFR high expression.
8. Evaluable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
9. Ability to swallow drugs.
10. Adequate organ function.
11. Voluntarily join the study and sign informed consent ad has good compliance.

Exclusion Criteria:

1. Prior therapies with EGFR targeted drugs including EGFR antibodies.
2. Previously treated with Irinotecan and Tegafur.
3. Anthracycline, nitrosourea, and mitomycin within 6 weeks; traditional Chinese medicine for anti-tumor within 2 weeks;immune anti-tumor therapy. within 8 weeks;other anti-tumor therapies within 4 weeks before randomization.
4. Not recovered from adverse events due to a previously administered agent.
5. Have undergone major surgery within 4 weeks prior to randomization (not including diagnostic surgery) or expect major surgery during the study period.
6. Previously or currently participating in other clinical trials within 4 weeks before randomization (subjects who have entered the follow-up period are calculated based on the last use of experimental drugs or devices).
7. Received a live vaccine within 28 days before randomization or plan to receive live vaccine after enrollment.
8. Received a strong inducer or inhibitor of CYP3A4 enzyme within 1 week or received Solivudine or its structurally similar drugs within 56 days prior to randomization.
9. Simultaneously receiving any other anti-tumor treatment.
10. Has a known additional malignancy previously within the last 5 years with the exception of basal cell carcinoma of the skin, squamous cell carcinoma of the skin or any other tumor that has been cured。
11. Central nervous system metastasis or uncontrolled central nervous system metastasis currently in need of treatment; or confirmed central nervous system metastasis, but not stable for more than 4 weeks after anti-tumor therapy; spinal cord compression, cancerous meningitis, or meningitis.
12. Clinically obvious gastrointestinal abnormalities, which may affect the intake, transport or absorption of drugs.
13. Having active gastrointestinal ulcer, active gastrointestinal bleeding, and perforation;
14. Risk of major bleeding or esophageal fistula;
15. Previous or present with interstitial lung disease or immunotherapy-associated pneumonia; currently suffering from drug-induced pneumonia, radiation pneumonitis requiring steroid therapy, or clinically symptomatic active pneumonia, or other moderate to severe lungs that seriously affect lung function disease
16. Active infection during the screening period (including but not limited to infection requiring intravenous drip therapy), or unexplained fever (> 38.5°C)within 2 weeks prior to randomization.
17. Has congenital or acquired immune deficiency (such as HIV infection).
18. Known active Hepatitis B or C.
19. Has any of the following diseases within the first 12 months of randomization: myocardial infarction, coronary artery bypass grafting or peripheral artery bypass graft surgery, heart failure (NYHA III to IV), etc and unstable angina with 6 months.
20. Has thrombosis or embolism occurred within the first 12 months of randomization, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis, pulmonary embolism with heparin or other similar drugs.
21. QTc interval (QTcF) corrected by Fridericia method> 470 ms; history of congenital long QT interval syndrome; any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation) Or torsion-type ventricular tachycardia); left ventricular ejection fraction (LVEF) <50%.
22. Allergies or contraindications to Z650 excipients (mannitol, sodium carboxymethyl starch, micronized silica gel, magnesium stearate, silicified microcrystalline cellulose), or to Irinotecan or Tegafur or its formulation ingredients.
23. Has uncontrolled pleural effusion, pericardial effusion, pelvic effusion, or ascites requiring repeated drainage.
24. Has a history of organ transplantation or a history of allogeneic bone marrow transplantation.
25. Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 6 months after the last dose of study medication.
26. Has other serious acute or chronic diseases and are not suitable for participating in clinical trials judged by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | up to approximately 22 months
  Defined as time from date of randomization to date of death due to any cause. OS was calculated using product-limit (Kaplan-Meier) method for censored data.

SECONDARY OUTCOMES:
Progression-free survival | up to approximately 22 months
  defined as the time from date of randomization until the earliest date of disease progression, as determined by independent central review of objective radiographic disease assessments per RECIST 1.1, or death from any cause, whichever comes first.
Objective response rate | up to approximately 22 months
  Objective response rate (ORR) is defined as the percentage of the participants in the analysis population who have a confirmed complete response (CR) or partial response (PR) based on RECIST 1.1 by investigators
Duration of response | up to approximately 22 months
  Defined as the time from the earliest date of qualifying response until earliest date of disease progression, per RECIST v1.1, or death from any cause, whichever comes first. Includes participants with complete response or partial response
Changes in health-related quality of life with esophageal cancer symptom scale | up to approximately 22 months
  To evaluate changes in health-related quality of life in patients with advanced esophageal cancer according to the Questionnaire
Incidence of Treatment-Emergent Adverse Events | up to approximately 22 months
  Assessed by Percentage of Participants With Adverse Events during the treatment assessed by NCI CTCAE 5.0
Apparent Oral Clearance (CL/F) of Lerotinib | up to approximately 22 months
  Defined as oral dose clearance
Apparent Volume of Distribution (Vd/F) of Lerotinib | up to approximately 22 months
  Apparent volume of distribution after administration.

CONTACTS AND LOCATIONS:
Overall Officials: JianMing Xu, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No